CLINICAL TRIAL: NCT02269358
Title: Phase 4, Open Lable Non Randomized un Controlled Study. Salvage Therapy With High/Low Methotrexate for Loss of Response to Infliximab Dose Escalation
Brief Title: Salvage Therapy With High/Low Methotrexate for Loss of Response to Infliximab Dose Escalation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and Nutrition unit., Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0143-14-WOMC
Record Dates: First submitted 2014-09-30; First posted 2014-10-21 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Addition of methotrexate (Experimental): Addition SC methotrexate at 15 mg/m2, not to exceed 25 mg/m2 . Patients in remission after 4 weeks will reduce their dose by halve. patients not in remission will continue the full dose until 12 weeks.
  Interventions: Drug: METHOTREXATE

INTERVENTIONS:
Drug: METHOTREXATE — Infliximab therapy after escalation. SC methotrexate at 15 mg/m2 , not to exceed 25 mg/m2 per week for 4 weeks. Patients in remission after 4 weeks reduce their dose by halve. patients not in remission will continue the full dose until 12 weeks.
  Other Names: Rheumatrex; Trexall

SUMMARY:
The goal of the present study is to evaluate if addition of methotrexate can restore remission after loss of response to infliximab after dose escalation.

another goal is to evaluate if low dose methotrexate can maintain remission achieved by regular dose methotrexate by 6 months.

DETAILED DESCRIPTION:
Background: IFX mono-therapy became the method of choice for treatment in pediatric CD, though this strategy has been called into question due to frequent loss of response to IFX requiring dose escalation of IFX or decreased intervals of IFX( up to 40% during the first year) (1). This loss of response has been attributed to development of ATIs and low trough levels of IFX, which can develop after the first infusions. This loss of response will often occur in patients with prior azathioprine exposure (2,3,4).

Currently , the first step during loss of response to infliximab in children is dose escalation either by decreasing the interval between infusions or doubling the dose. However, patients with persistent antibodies or high titers are likely to fail even with dose escalation. The Sonic trial clearly demonstrated that combination therapy with a thiopurine may be more effective than Anti TNF alpha monotherapy (2). Ben Horin et al demonstrated that antidrug antibodies can be reversed and improved anti TNF trough levels obtained by adding an immunomodulator to failed monotherapy due to an antidrug antibody (3).

We have previously shown that in patients with a previous loss of response to two biologics leading to cessation of both biologics can respond to reinduction with adalimumab and methotrexate . Among 12 patients (10 children and two adults) , 6 obtained complete remission. We subsequently lowered the does in several patients without loss of response, and tried stopping methotrexate in 3 patients. All 3 patients relapsed within months of complete cessation of methorexate.In this previous study we took two separate actions that restored response, re-induction and methotrexate therapy. In the current proposal we will take patients that are on escalated therapy and just add methotrexate, in order to evaluate if adding methotrexate once weekly can restore response after loss of response to infliximab after failed dose escalation.It is important to note that methotrexate does not increase the risk of malignancy as co-therapy as far as we know.

Methods: It is a prospective open label phase 4, non randomized uncontrolled study in a small cohort of patients to evaluate if addition of methotrexate can restore remission after loss of response to infliximab after dose escalation in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Established diagnosis of Crohns disease.
3. Age: 8 - 18 years ( inclusive)
4. Active disease PCDAI >10 at least two weeks after infusion.
5. On Infliximab with at least 3 prior infusions, and still active despite a decreased dose interval ( ≤ 6 weeks) or increased dose of infliximab (≥7.5 mg/kg /dose q 8 weeks).

Comment: Patients who are on combination therapy with a stable thiopurine>8 weeks can also be included ( thiopurine will be stopped at enrollment).

-

Exclusion Criteria:

1. Patients who are primary non responders after first two doses 2. Patients who have had to stop infliximab due to side effects. 3. Patients with known intolerance to methotrexate. 4. Elevated ALT >1.5 normal. 5. Pregnancy. 6. Patients who have insulin-dependent diabetes 7. Patients who have significantly impaired renal function 8. Current bacterial infection/ inflammation including Hepatitis B or C and Pneumonia.

-

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2015-07; Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
remission | at 12 weeks
  remission without additional therapy.

SECONDARY OUTCOMES:
Remission | 6 months
Trough levels | week 12
ATIs | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Study Chair — Pediatric Gastroenterology and Nutrition Unit, The E. Wolfson MC, Tel-Aviv University, Holon, Israel
Locations (1):
- The E. Wolfson.Medical Center, Holon, Israel